CLINICAL TRIAL: NCT06379984
Title: Rapid Outpatient Low-dose Initiation of Buprenorphine for Individuals With OUD Using Fentanyl
Brief Title: Rapid Outpatient Low-dose Initiation of Buprenorphine for OUD With Fentanyl Use
Acronym: ROLDI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kyle Kampman, Professor of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 855013
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use Disorder
Keywords: Fentanyl; Buprenorphine; Low-dose initiation; Opioid addiction; Opiate
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rapid outpatient low-dose initiation (Experimental): Participants randomized to low-dose initiation will be instructed to arrive to the research unit without withdrawal. Participants with COWS <4 will be admitted to the research unit to begin induction. They will be administered 0.5, 0.5, 1, 1, 1, 4, and then 8 mg as sublingual buprenorphine films with doses scheduled every 2 hours. They will then continue 8mg twice daily (or up to three times daily) as maintenance treatment.
  Interventions: Drug: Buprenorphine
- Standard initiation (Active Comparator): Participants randomized to standard induction will be instructed to arrive to the research unit with mild withdrawal and to have abstained from opioids for at least 8 hours, per ASAM Guidelines. Participants with COWS 4 or higher on initial assessment will be admitted to the research unit to begin induction.
  Standard initiation will follow guidelines from the 2020 Focused Update of the ASAM National Practice Guidelines. Once participants have had at least 8 hours of abstinence and have reached COWS 11 or greater, they will be given 2 mg sublingual buprenorphine, followed 2 hours later by 2 mg, followed 2 hours later by 4 mg, followed 2 hours later by 8 mg. They will then continue 8 mg twice (or up to three times) daily as maintenance treatment.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Sublingual buprenorphine

SUMMARY:
The goal of this clinical trial is to learn if buprenorphine can be started for opioid use disorder with fentanyl use without requiring or precipitating opioid withdrawal. To be eligible, participants must have moderate or severe opioid use disorder and must have fentanyl detected on a urine drug test.

Participants will be admitted to a monitored research unit for the trial. They will be randomized to start buprenorphine with either standard initiation or with a new approach called rapid outpatient low-dose initiation (ROLDI).

For standard initiation, participants will be instructed to arrive to the unit with at least 8 hours since last fentanyl use. Once they have at least moderately severe opioid withdrawal (Clinical Opiate Withdrawal Scale [COWS] 11 or higher), participants will receive 2 mg, 2 mg, 4 mg, and then 8 mg sublingual buprenorphine, with doses every 2 hours. They will then continue 8 mg twice daily (or up to three times daily). This is the current standard of care.

For ROLDI, participants will not be required to have a period abstinence, they will have no or minimal withdrawal (COWS 4 or less) when starting buprenorphine, and participants will take 0.5 mg, 0.5 mg, 1 mg, 1 mg, 1 mg, and then 4 mg sublingual buprenorphine with dosing every two hours. They will then continue 8mg twice daily (or up to three times daily).

The main aim of this clinical trial is to assess whether ROLDI is safe, feasible, acceptable to patients, and worthwhile to study in a larger trial. The secondary aim is to describe fentanyl and norfentanyl pharmacokinetics (that is to say, fentanyl and norfentanyl concentration in blood and urine) during early abstinence to understand why some people using fentanyl develop precipitated withdrawal with standard initiation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older
* Male, female, transgender, or non-binary
* DSM-5 criteria for opioid use disorder, moderate to severe
* Fentanyl positive on urine drug test
* Able to provide written informed consent in English prior to any study-related procedure

Exclusion Criteria:

* Pregnancy or actively lactating
* Previously documented hypersensitivity or allergy to buprenorphine or naloxone
* DSM-5 criteria for substance use disorder other than opioid use disorder (e.g., cannabis, cocaine, alcohol)
* Current benzodiazepine use
* Urine drug testing at screening positive for buprenorphine and/or methadone
* AST and/or ALT >3x upper limit of normal or total bilirubin >1.5x upper limit of normal
* eGFR <30 mL/min
* Use of CYP3A4-metabolized agents such as azole antifungals, macrolides, and protease inhibitors
* High risk of severe medetomidine withdrawal based on drug urine testing for medetomidine, prior withdrawal syndrome requiring intensive care unit admission, and/or patient-reported severe nausea/vomiting during early withdrawal, at the discretion of the study physicians.
* Significant medical symptoms (e.g. severe respiratory insufficiency), psychiatric symptoms, or dementia that, in the opinion of the investigators, would preclude compliance with the protocol, cooperation in the study, obtaining informed consent, or ability to safely participate in the study
* Pending legal action that could prohibit participation and/or compliance in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Initiation of buprenorphine maintenance without precipitated withdrawal | 10 hours
  The proportion of subjects who complete buprenorphine initiation without precipitated withdrawal. Completing buprenorphine initiation is defined as reaching 8mg or more total daily dose of sublingual buprenorphine without termination of buprenorphine initiation for any reason. Precipitated withdrawal is defined as an increase in COWS of 6 or more (compared to the COWS immediately preceding the most recent dose of buprenorphine) within 2 hours of the most recent dose of sublingual buprenorphine.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No